CLINICAL TRIAL: NCT04933591
Title: Impact of Treatment With VENARUS® on Vein-specific by Determining the Level of Monocyte Chemoattractant Protein 1 in Varicose Veins Blood
Brief Title: Impact of Treatment With VENARUS® on the Level of Monocyte Chemoattractant Protein 1 in Varicose Veins Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Igor Zolotukhin, Professor, Pirogov Russian National Research Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NIS-ВЕН-19.03
Record Dates: First submitted 2021-06-07; First posted 2021-06-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — Diosmin; Hesperidin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Individuals aged 18-50 with varicose veins and CEAP C2-C4, Ep, As, Pr. Clinical and ultrasound examinations will be used to confirm varicose veins disease. It is planned to take blood samples from a varicose vein before and after administration of Venarus® (100 mg hesperidin + 900 mg diosmin) for 2 months
  Interventions: Drug: Diosmin / Hesperidin
- control group (No Intervention): Individuals aged 18-50 with varicose veins and CEAP C2-C4, Ep, As, Pr vein. Clinical and ultrasound examinations will be used to confirm varicose veins disease. It is planned to take blood samples from a varicose vein at inclusion and 2 months later/

INTERVENTIONS:
Drug: Diosmin / Hesperidin — Venoactive drugs are used for patients with varicose veins as a tool for alleviating symptoms
  Other Names: Venoactive drug
  Arms: study group

SUMMARY:
This study is designed to find if the venoactive drug contained diosmin and hesperidin is able to work against chronic vein-specific inflammation by changing the level of Monocyte Chemoattractant Protein 1. This chemokine is involved in the vein wall remodeling in patients with lower limb varicose veins.

DETAILED DESCRIPTION:
The study is a post-registration open-label observational prospective single-center study with minimal intervention. Individuals aged 18-50 with varicose veins and CEAP C2-C4, Ep, As, Pr will be invited to participate in the study.

Those who agree, will be examined both clinically and by duplex ultrasound. Medical history of participants will be taken, demographic data will be collected. Blood will be drawn from the varicose vein of the affected limb. Discomfort in the affected limb will be evaluated by a visual-analog scale. Duplex ultrasound will be used in every resident to reveal pathological venous reflux in deep and superficial veins.

ELIGIBILITY:
Inclusion Criteria:

* • both female and male

  * age from 18 to 50 years old
  * Verified diagnosis of chronic venous insufficiency CEAP C2-C4
  * signed infromed consent
  * Absence of any other treatment 2 weeks before the start of the study and throughout the duration of the study

Exclusion Criteria:

* • age less than 18 and more than 50 years

  * Previously performed invasive interventions for varicose veins on any of the lower extremities
  * No visible varicose veins
  * Thrombophlebitis and deep vein thrombosis of the lower extremities in the past
  * Taking prohibited pre-trial therapy
  * Contraindications to taking Venarus®
  * not signed informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the level of Monocyte Chemoattractant Protein 1 level in blood taken from varocse vein | 2 months
  Blood samples will be taken from varicose veins and level of cytokine Monocyte Chemoattractant Protein 1 will be measured by immunofluorescence. After 2 months measurement will be repeated and the change will be registered.

SECONDARY OUTCOMES:
Change from baseline of discomfort related to symptoms of varicose veins (i.e., pain, heaviness, etc.) | 2 months
  Discomfort will be measured by visual-analogue scale. After 2 months measurement will be repeated and the change will be registered.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Zolotukhin, PhD, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- Pirogov Russian National Research Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No